CLINICAL TRIAL: NCT02429453
Title: Fresh Frozen Plasma Versus Four Factor Prothrombin Complex Concentrate for Reversal of Vitamin K Antagonists in Intracranial Hemorrhage
Brief Title: FFP Versus PCC in Intracranial Hemorrhage
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of enrolment
Sponsor: University of Utah (Other)
Responsible Party: Principal Investigator, Jian Guan, Neurosurgery Resident, University of Utah
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB_00078143
Record Dates: First submitted 2015-04-21; First posted 2015-04-29 (Estimated); Last update posted 2016-11-16 (Estimated); Status verified 2016-11

CONDITIONS: Intracranial Hemorrhage, Traumatic; Intracranial Hemorrhage, Spontaneous
Keywords: Warfarin; Traumatic intracranial hemorrhage; prothrombin complex concentrate; fresh frozen plasma; Spontaneous intracranial hemorrhage
MeSH Terms: conditions — Intracranial Hemorrhage, Traumatic; Intracranial Hemorrhages; Hemophilia B

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Fresh Frozen Plasma (Active Comparator): Administration of a single dose of fresh frozen plasma based on INR per the following regimen: 2U for INR of 2-2.5; 3U for INR of 2.5-3; 4U for INR of 3-3.5; 5U for INR of 3.5-4; 6U for INR of 4+
  Interventions: Biological: Fresh Frozen Plasma
- Four Factor Prothrombin Complex Concentrate (Experimental): Administration of a single dose of four factor prothrombin complex concentrate per the following dosing regimen: 25 U/kg for INR of 2-4; 35 U/kg for INR of 4-6; 50 U/kg for INR of 6+; maximum dosing weight of 100kg, patients may be dispensed +/- 10% of ordered dose
  Interventions: Drug: Four Factor Prothrombin Complex Concentrate

INTERVENTIONS:
Drug: Four Factor Prothrombin Complex Concentrate — A purified, non-activated prothrombin complex concentrate containing factors II, VII, IX and X and proteins C & S
  Other Names: Kcentra
  Arms: Four Factor Prothrombin Complex Concentrate
Biological: Fresh Frozen Plasma — A pooled collection of plasma from donors
  Arms: Fresh Frozen Plasma

SUMMARY:
The goal of this study will be to determine whether PCC confers any benefits over FFP in traumatic and spontaneous intracranial hemorrhage with respect to multiple factors including time to correction, absolute international normalized ratio correction amount, cost, need for surgical intervention, and radiographic bleed expansion through a prospective, randomized control trial.

DETAILED DESCRIPTION:
Vitamin K antagonists in general and Coumadin in particular remains the most common form of outpatient anticoagulation in patients today. Despite the therapeutic benefits of these agents, bleeding in general and intracranial bleeding in particular are significant risks associated with these medications. Intracranial bleeding on oral anticoagulation agents are associated with a 20% increase in 30 day mortality versus non-anticoagulated controls, and rapid reversal of vitamin K antagonists in this population has been shown to have survival benefits.

Historically, vitamin K antagonists have been reversed using fresh frozen plasma (FFP) transfusions which, though effective, often incur delays due to the time required to obtain a type & screen, thaw the product, and administer the product to the patient. In 2013, the FDA approved 4-factor prothrombin complex (PCC), a concentrate of factors II, VII, IX, X, protein C and protein S for use as a method for correcting vitamin K antagonist related coagulopathy. Though large, prospective randomized control trials have demonstrated efficacy and safety in a general population of all-comers bleeding, there is very little literature regarding the benefits of PCC versus FFP in the traumatic and spontaneous intracranial hemorrhage population.

Current standard of care in patients with traumatic and spontaneous intracranial hemorrhage who are on vitamin K antagonists is to reverse the effect of these agents with FFP or PCC. The choice of which agent to use is currently determined by both availability of each agent and surgeon preference. For this study, there will be an equal likelihood of either treatment being given.

The goal of this study will be to determine whether PCC confers any benefits over FFP in traumatic and spontaneous intracranial hemorrhage with respect to multiple factors including time to correction, absolute international normalized ratio correction amount, cost, need for surgical intervention, and radiographic bleed expansion through a prospective, randomized control trial.

ELIGIBILITY:
Inclusion Criteria:

* Coumadin use
* INR of 2.0 or higher on arrival at the study center
* Evidence on cranial imaging of spontaneous intracranial hemorrhage, subdural hematoma, epidural hematoma, cerebral contusion, traumatic subarachnoid hemorrhage, or traumatic intraparenchymal hemorrhage

Exclusion Criteria:

* Unable to obtain consent
* Estimated survival <24 hours
* Hypersensitivity to 4 factor prothrombin complex concentrate
* Concomitant use of novel vitamin K antagonists
* Religious/social prohibition to receiving blood products
* Need for emergent, non-neurosurgical operative intervention
* Mechanical heart valves

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-04; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Rapid reversal of warfarin as measured by international normalized ratio (INR) drawn at 30 minutes after transfusion | 30 minutes after transfusion completion
  INR level 30 minutes after transfusion completion of FFP or 4 factor prothrombin complex concentrate

SECONDARY OUTCOMES:
Radiographic expansion of traumatic intracerebral hemorrhage as measured by CT scan within 24 hours of presentation | 24 hours after presentation
  Expansion of blood on repeat CT scan of >10%
Timing of reversal of warfarin as measured by INR drawn at 3 hours, 8 hours and 24 hours after transfusion | 3-24 hours after completion of FFP or 4 factor prothrombin complex concentrate transfusion
  INR level at 3 hours, 8 hours and 24 hours after transfusion completion of FFP or prothrombin complex concentrate
Thromboelastography response as measured by results of ROTEM analysis at 30 minutes and 24 hours after transfusion | 30 minutes and 24 hours after completion of FFP or 4 factor prothrombin complex concentrate transfusion
  Results of ROTEM analysis at 30 minutes and 24 hours after transfusion
Absolute INR reversal as measured by INR drawn 24 hours after transfusion | 24 hours after completion of FFP or 4 factor prothrombin complex concentrate transfusion
  Difference between initial INR and INR 24 hours after completion of transfusion
Need for operative intervention as measured by need for neurosurgical procedure during the hospitalization | During duration of hospital stay, an expected average of 1 week
  Need for operative intervention during hospitalization related to initial trauma
Estimated blood loss during any neurosurgical procedure | During duration of hospital stay, an expected average of 1 week
  Estimated blood loss during any neurosurgical interventions during the hospitalization
Further transfusion needs as measured by number of units of blood/platelet/plasma products transfused during the hospitalization | During duration of hospital stay, an expected average of 1 week
  Need for blood product transfusions during hospitalization
In hospital mortality | During duration of hospital stay, an expected average of 1 week
  Mortality during hospital stay
Total hospital cost | During duration of hospital stay, an expected average of 1 week
  Total cost of hospital stay based on hospital charges
30 day outcome as measured by the Glasgow outcome score | 30 days after discharge
  Glasgow outcome score 30 days after discharge
Complications as measured by development of deep vein thrombosis, pulmonary embolism, myocardial infarction, stroke, unanticipated intubation, heart failure, or need for aggressive diuresis during the hospitalization | During duration of hospital stay, an expected average of 1 week
  Development of deep vein thrombosis, pulmonary embolism, myocardial infarction, stroke, unanticipated intubation, heart failure, or need for aggressive diuresis

CONTACTS AND LOCATIONS:
Locations (1):
- University of Utah Medical Center, Salt Lake City, Utah, United States

REFERENCES:
- [Derived] Eilertsen H, Menon CS, Law ZK, Chen C, Bath PM, Steiner T, Desborough MJ, Sandset EC, Sprigg N, Al-Shahi Salman R. Haemostatic therapies for stroke due to acute, spontaneous intracerebral haemorrhage. Cochrane Database Syst Rev. 2023 Oct 23;10(10):CD005951. doi: 10.1002/14651858.CD005951.pub5. PMID 37870112